CLINICAL TRIAL: NCT00455169
Title: Influenza Vaccine Immunogenicity in Extremely Premature Infants
Brief Title: Influenza Vaccine in Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Thrasher Research Fund (Other); University of Miami (Other); Wake Forest University Health Sciences (Other); State University of New York at Buffalo (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Professor, University of Rochester
Other Study IDs: URRSRB15397A
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Influenza; Infant, Premature
Keywords: Influenza; Infant, Premature; Immunization; Vaccination
MeSH Terms: conditions — Influenza, Human; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No retention
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Premature infants
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine
- 2: Full term infants
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza Vaccine — Influenza vaccine

SUMMARY:
Background. Influenza is increasingly recognized as causing severe respiratory illness in children. High-risk infants, like former premature infants, and particularly those with lung disease, have influenza hospitalization rates about five times higher than healthy children. Influenza vaccine does not protect young children against influenza as well as it does healthy adults. A small study that measured antibodies (proteins that protect against infection) to influenza suggested that premature infants get even less protection from influenza vaccine than full-term infants. More information about influenza vaccine in premature infants is needed. The overall goals of this project are to collect information about the how well the influenza vaccine induces antibody production, and to develop the collaborative network of centers necessary for a larger trial of influenza vaccine in premature infants.

Objective and Hypotheses. The objective of this study is to measure the amount of protective antibody produced by influenza vaccine in premature (less than 30 weeks' [about 7 months] gestation at birth), extremely-low-birth-weight (1000 grams [2¼ pounds] or less at birth) infants. Influenza vaccine needs to be given yearly. We will assess premature infants during their first series of influenza vaccines. We hypothesize that the levels of antibody will be lower in premature infants receiving their first series of influenza vaccine than in full-term infants.

Design. We will measure the immune response in premature and full term infants. During the 2007-2008 influenza season, a total of 92 subjects, divided among 2 groups (premature infants 6-17 months old receiving their first influenza vaccine series and full-term infants 6-17 months old receiving their first influenza vaccine series) will be recruited at a consortium of five centers (the University of Rochester, the University of Texas Southwestern Medical Center, Wake Forest University, the University of Miami and the State University of New York at Buffalo), receive 2 doses of influenza vaccine, and have antibody and immune cell responses to each vaccine component measured 4-6 weeks after the second dose of vaccine.

Potential Impact. If this study and future investigations suggested ways to improve premature infants influenza vaccine responses, they could lead to changes in recommendations for the number or timing of vaccine doses or of the type of vaccine used in this high-risk group.

DETAILED DESCRIPTION:
Background. Influenza infection causes an estimated 1 million deaths worldwide yearly. Severe influenza respiratory disease is increasingly recognized in children. Influenza hospitalization rates in high-risk infants, such as premature infants, are increased some five-fold over rates in other children. Influenza vaccine immunogenicity is generally modest even in healthy children, and influenza vaccines have been incompletely studied in premature infants. Further investigation is required to optimize vaccine responses in premature infants. The overall goals of this project are to generate estimates of effect size and variance of influenza vaccine immunogenicity for use in planning a larger multi-center trial, and to develop the collaborative network of centers necessary for such a trial.

Objective and Hypotheses. The primary objective of this study is to measure influenza vaccine immunogenicity in extremely-low-birth-weight (ELBW, < 1001 grams at birth), premature (< 30 weeks' gestation) infants receiving trivalent, inactivated, split-virion influenza vaccine (TIV). We hypothesize that the geometric mean titer (GMT) of antibody to each of the three vaccine components will be lower in ELBW infants receiving their first series of TIV than in full-term (FT, >37 weeks' gestation), normal-birth-weight (>2500 grams) infants.

Specific Aim. To measure the humoral and cellular immunogenicity of influenza vaccine in extremely-low-birth-weight (ELBW, greater than or equal to 1000 grams at birth), premature infants receiving trivalent, inactivated, split-virion influenza vaccine (TIV) for their first influenza vaccine series in 2007-8.

Design. This prospective, cohort, immunogenicity study will estimate the GMT to influenza in ELBW infants, with a comparison group of FT infants. Using the established vaccine study infrastructure at a consortium of five centers (the University of Rochester, the University of Texas Southwestern Medical Center, Wake Forest University, the University of Miami and the State University of New York at Buffalo), we will recruit 46 un-immunized (for influenza) ELBW infants, 6-17 months old and 46 un-immunized FT infants, 6-17 months old. Infants will receive the recommended 2 doses of TIV, 4 weeks apart, with blood drawing at the first vaccine dose and 4-6 weeks after the second. Antibody to each vaccine component will be measured by hemagglutination inhibition. The frequency of hemagglutinin-specific T cell interleukin (IL)-2, IL-4 and interferon gamma (IFNγ) responses will be measured by ELISPOT assay. The primary outcome will be influenza GMT. A sample size of 46 subjects per group provides 80% power, using a two-sided alpha = 0.05, to detect a 1.5-fold difference in GMT between groups, assuming a standard deviation (SD) spanning 0.5 to 2.0 times the value of each GMT. In addition, the five-center consortium will monitor the quality of the collaboration, strengthen its capabilities through the design and implementation of a secure, web-based information system, and expand its efforts by seeking additional, outside funding to implement a companion protocol assessing live attenuated influenza vaccine in premature infants.

Potential Impact. This study is designed to assess the immunogenicity of the current generation of influenza vaccines in premature infants. This and future trials assessing novel immunization strategies (such as an additional vaccine dose) or vaccines (for instance, the live attenuated influenza virus vaccine) in premature infants could eventually lead to the tailoring of specific vaccine strategies for this high-risk group. In addition, this proposal would bring to maturity a multi-center, collaborative mechanism for vaccine trials in premature infants.

ELIGIBILITY:
Inclusion criteria. Subjects must meet all relevant criteria to participate.

1. (a) Former premature (< 30 weeks' gestation at birth), ELBW (<1001 grams' birth weight) infant, 6 months, 0 days - 17 months, 31 days of age., OR (b) Former full term (37-42 weeks' gestation at birth), normal birth weight (>2500 grams' birth weight) infant, 6 months, 0 days - 17 months, 31 days of age.
2. No prior influenza immunization.
3. Eligible for influenza immunization.
4. Parental permission.
5. Agreement of primary care provider.
6. Parents likely to be able to comply with study visits.

Exclusion criteria. Subjects may not participate if they meet any one of these criteria.

1. Known immunodeficiency.
2. Systemic corticosteroid administration at time of study enrollment.
3. Requiring supplemental oxygen.
4. Contraindication to influenza immunization (e.g. egg allergy).
5. Physician-diagnosed influenza illness in the current influenza season.
6. Any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the subject.

Ages: 6 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants < 30 week's gestation, < 1001 grams' birth weight or full-term infants 37-42 week's gestation >2500 grams' birth weight
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl T D'Angio, MD, Principal Investigator — University of Rochester
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - State University of New York at Buffalo, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] D'Angio CT, Heyne RJ, Duara S, Holmes LC, O'Shea TM, Wang H, Wang D, Sanchez PJ, Welliver RC, Ryan RM, Schnabel KC, Hall CB; Premature Infant Vaccine Collaborative. Immunogenicity of trivalent influenza vaccine in extremely low-birth-weight, premature versus term infants. Pediatr Infect Dis J. 2011 Jul;30(7):570-4. doi: 10.1097/INF.0b013e31820c1fdf. PMID 21273938